CLINICAL TRIAL: NCT03576417
Title: A Phase III Randomized Trial of Post-operative Adjuvant Nivolumab and Concomitant Chemo-radiotherapy in High-risk Patients With Resected Squamous Cell Carcinoma of Head and Neck
Brief Title: A Trial Evaluating the Addition of Nivolumab to Cisplatin-RT for Treatment of Cancers of the Head and Neck
Acronym: NIVOPOSTOP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: For Drug Consulting (Other); Eurofins (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2018-01
Record Dates: First submitted 2018-06-01; First posted 2018-07-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RT+ cisplatin (Active Comparator): 100 mg/m2 of cisplatin on days 1, 22,43 of RT
  Interventions: Drug: Cisplatin; Radiation: RT
- RT+ cisplatin + nivolumab (Experimental): * 240 mg of nivolumab 3 weeks before RT-Cisplatin
  * 360 mg of nivolumab on days 1, 22,43 of -RT-cisplatin
  * 480 mg of nivolumab for maintenance
  Interventions: Drug: Cisplatin; Drug: Nivolumab; Radiation: RT

INTERVENTIONS:
Drug: Cisplatin — Intravenous
Drug: Nivolumab — Intravenous
  Arms: RT+ cisplatin + nivolumab
Radiation: RT — IMRT 66 Gy / 6.5 weeks
  Other Names: IMRT

SUMMARY:
The purpose of this study is to determine the efficacy of nivolumab + cisplatin-RT relative to standard of care (SOC) cisplatin-RT alone, using the disease-free survival (DFS by investigator imaging assessment) as primary endpoint )

DETAILED DESCRIPTION:
This open-label, randomized, controlled, multicenter phase III study will include 680 patients who have been operated for their LA SCCHN and exhibiting extra capsular extension (ECE) and/or positive margins (high risk). Subjects will be randomized (1:1) to receive post-operative concomitant cisplatin-RT with or without nivolumab.

The study is designed with the general objective of demonstrating that treatment with nivolumab in combination with 3 cycles of cisplatin during RT is more efficient and not more toxic than the SOC 3 cycles of cisplatin during RT.

Stratification will be based on the P16 status (immunohistochemistry assay on surgical sample). Two classes: Oropharyngeal Cancer (OPC) p16 positive versus OPC p16 negative or not OPC.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 75 years
2. Performance Status (PS) ECOG 0-1 (Appendix 2)
3. Written informed consent
4. Recording of alcohol consumption and smoking history
5. Histologically proven squamous cell carcinoma of the head and neck from one or more of the following primary sites: oral cavity, oropharynx, hypopharynx or larynx
6. Squamous cell carcinoma of the head and neck treated by primary surgery
7. Histopathological classification: pStage III or IV. However, Oropharyngeal Cancer pStage II p16 positive with pT3N1 or pT4N1 and tobacco consumption ≥20 packs/year are eligible. (American Joint Committee on Cancer 8th edition)
8. Subject must have complete macroscopic resection.
9. Subject must be free of disease
10. Recovery from the surgical procedure allowing for cisplatin-Radiotherapy
11. Radiotherapy planned to start within 4 to 9 weeks after surgery. However, a maximum of 1 additional week could be considered in case of delay due to healing or logistical problem
12. Patient/tumor carrying a high risk of relapse with:

    * Extra-capsular extension (ECE),
    * Multiple peri-neural invasion
    * Multiple nodal extension without ECE (≥ 4 nodes)
    * Positive margins (R1 or close margin ≤ 1 mm) R1 is microscopic residual disease and close margin is R0 with a minimum margin ≤ 1 mm in any direction.
13. Adequate tumor specimen from archived or resected tissue available for PD-L1, TILs and immune landscape and other biomarker evaluation
14. For oropharyngeal tumor, known p16 status (by IHC)
15. Patient's ability to receive cisplatin 100 mg/m2 for 3 cycles:

    * Creatinine Cclearance (CrCl) ≥ 60 mL/min (measured or calculated by Cockcroft and Gault method) or estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73m2 (determined by CKDEPI or MDRD method). The highest value should be considered if both are assessed.
    * Absolute neutrophil count ≥1 500/mm3, platelets ≥100 000/mm3, haemoglobin ≥ 9 g/dL, aspartate transaminase (AST) and alanine transaminase (ALT) less than 2.5 times the upper limit of the normal range (ULN), total bilirubin ≤ 1.5 mg/dL(except Gilbert Syndrom: < 3.0 mg/dL).
    * Peripheral neuropathy ≤ grade 1
    * No hearing loss (assessed clinically and confirmed by audiogram if doubtful)
    * Cardiac function compatible with hyperhydration
    * No administration of prophylactic phenytoin
    * Patients aged 71-74 years,must be fit according to geriatric evaluation

Exclusion Criteria:

1. Nasopharyngeal, paranasal sinuses, nasal cavity tumours or thyroid cancers
2. Squamous cell carcinoma involving cervical neck nodes with unknown primary site
3. Metastatic disease
4. Incomplete macroscopic resection (R2), as stated in the surgical report
5. Known active viral infection Human Immunodeficiency Virus (HIV), Hepatitis B/C) or known history of positive test for HIV, active autoimmune disease and/or an active immunodeficiency or ongoing immunosuppressive therapy
6. Active Central Nervous System disease
7. Interstitial lung disease
8. Active infection
9. Any prior treatment for the current head and neck cancer other than primary surgery. This will include but is not limited to: prior tyrosine kinase inhibitors, any monoclonal antibody, induction chemotherapy, prior RT, or use of any investigational agent
10. Concurrent treatment with any other systemic anti-cancer therapy that is not specified in the protocol
11. Concomitant treatment with any drug on the prohibited medication list such as live vaccines. Live vaccines administered more than 30 days before study entry are permitted
12. History of other malignancy within the last 3 years (exception of in situ carcinoma, thyroid papillary carcinoma, skin carcinomas, localized prostate carcinoma Gleason 6 and in situ breast carcinoma)
13. Pregnant, breastfeeding patients, and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in the protocol for the duration of the study and for at least 6 months after the last dose of cisplatin and 5 months after the last dose of nivolumab
14. Male patients who are unwilling or unable to use contraception methods for the duration of the study and for at least 6 months after the last dose of cisplatin.
15. Severe acute or chronic medical conditions including colitis, pneumonitis, pulmonary fibrosis, laboratory abnormalities or other significant disease which, in the judgment of the investigator, as a result of the medical interview, physical examinations, or screening investigations would make the patient inappropriate for entry into the trial
16. Known hypersensitivity to study drugs
17. Prior organ transplantation including allogenic stem-cell transplantation
18. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
19. Concurrent enrolment in another clinical trial using an investigational anti-cancer treatment within 28 days prior to the first dose of study treatment
20. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
21. Any psychiatric condition (including active suicidal ideation), or psychological, or familial, or sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
22. Individuals deprived of liberty or placed under the authority of a tutor.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years after the end of RT
  The time between the date of randomization and the date of first loco-regional or distant recurrence or death (of any cause) whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 60 months after the end of treatment
  Time between the date of randomization and death
Acute toxicity | During treatment and until 90 months after the end of RT
  The maximal grade of each toxicity observed during radiotherapy plus concomitant treatment graded according to the NCI CTCAE v5.0
Late toxicity | 1 to 5 years after radiotherapy
  Late toxicity from 1 year to 5 years after radiotherapy will be categorized in three categories (none, grade 1-2, or grade 3-4), and compared between the two arms using generalised linear models for multinomial variables with a cumulative logit link

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Bourhis J, Auperin A, Borel C, Lefebvre G, Racadot S, Geoffrois L, Sun XS, Saada E, Cirauqui B, Rutkowski T, Henry S, Modesto A, Johnson A, Chapet S, Calderon B, Sire C, Malard O, Bainaud M, Da Silva Motta A, Thureau S, Pointreau Y, Blanchard P, Buiret G, Bozec L, Lopez S, Vanbockstael J, Bosset M, Greilsamer C, Daste A, Bruna A, N'Guyen F, Plana M, Iruarrizaga E, Temam S, Even C, Ruiz EP, Bert M, Karamouza E, Thariat J, Kazmierska J, Psyrri A, Mesia R, Tao Y. Nivolumab added to cisplatin and radiotherapy versus cisplatin and radiotherapy alone after surgery for people with squamous cell carcinoma of the head and neck at a high risk of relapse (GORTEC 2018-01 NIVOPOST-OP): a randomised, open-label, phase 3 trial. Lancet. 2026 Jan 24;407(10526):363-374. doi: 10.1016/S0140-6736(25)01850-1. Epub 2025 Dec 22. PMID 41448222